CLINICAL TRIAL: NCT03785158
Title: Melatonin for Preventing Postoperative Delirium in Elderly Patients; a Multi-centre Randomized Placebo Controlled Pilot Study
Brief Title: MIND After Surgery
Acronym: MIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 5506
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-07

CONDITIONS: Post-operative Delirium; Major Non-cardiac Surgery
Keywords: Delirium; Elderly patients having non-cardiac surgery; Melatonin; sleep quality; sleep deprivation; sleep-wake cycle
MeSH Terms: conditions — Emergence Delirium; Delirium; Sleep Initiation and Maintenance Disorders; Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: This is a randomised, placebo-controlled, two arm parallel design pilot RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Active Comparator): 3 mg of liquid melatonin by oral route for 8 days. The 1st dose will be given 1-2 hours prior to the surgery, followed by bed time doses (between 7-9 pm) given on postoperative day (POD) 1 until discharge or for the first 7 days.
  Interventions: Other: Liquid Melatonin
- Placebo Group (Placebo Comparator): Similar looking/tasting 3 mg (5 ml) placebo syrup administered preoperatively by oral route and for the next 7 days or until discharge. The 1st dose will be given 1-2 hours prior to the surgery, followed by bed time doses (between 7-9 pm) given on postoperative day (POD) 1 until discharge or for the first 7 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Liquid Melatonin — Melatonin is a natural supplement.
  Arms: Melatonin
Other: Placebo — Similar looking/tasting placebo syrup
  Arms: Placebo Group

SUMMARY:
Delirium is the most common neurological adverse outcome in elderly surgical patients. It is associated with an increased mortality and morbidity, including need for prolonged hospital stay and institutional care. Despite this, there are no effective preventive strategies. Melatonin is a hormone released from the pineal gland. It is used to improve sleep quality and to treat jet lag. Small studies have suggested that it can decrease the chances of delirium. Since the existing literature is small and uncertain, it is important to test its benefit in a large sample to help guide clinicians. This proposed trial is aimed at testing assessing the feasibility of a large, multi-center, randomized control trial to decrease the incidence of postoperative delirium.

DETAILED DESCRIPTION:
Delirium is defined as an acute and fluctuating disturbance in cognition characterized by alterations in the level of attention and awareness, which develops over a relative short period of time and represents a change from the subject's baseline. Its incidence increases with age and occurs in nearly 50% of elderly inpatients. Postoperative delirium (POD) increases the risk of patient morbidity and mortality and thereby increasing the cost for the health care system. Increased risk of mortality persists even three years after hospitalization, and is an independent risk factor for urinary incontinence, falls, and decubitus ulcers.

A large prospective study of 1341 patients having non-cardiac surgery with a postoperative stay of at least 48 hours, reported an overall incidence of 9% in >50 years and 15% in >70 years. Another recent study involving 566 patients of similar surgical cohort reported an incidence of 24%.

With no current effective treatment, there is a greater focus on prevention of delirium. Approximately 15% of all POD could be preventable. Preventive strategies can be pharmacological and non-pharmacological. Non-pharmacological strategies are multifaceted and involve different interventions. Among attempted pharmacological options, none have really shown much promise and many suffer from associated adverse effects.

Melatonin is a pineal gland hormone that regulates the sleep-wake rhythm. Disruption of the sleep-wake cycle is observed in delirium. Abnormal tryptophan metabolism is hypothesized as a cause for delirium and melatonin supplementation is observed to decrease the breakdown of tryptophan and serotonin through positive feedback. In patients who develop POD, low tryptophan and serum melatonin levels were observed. Other advantages of melatonin, being a natural supplement, include improved sleep, sparing of sedatives, minimal potential for abuse, or hangover effects.

Systematic reviews done with the existing literature specific to melatonin by a literature search of MEDLINE, EMBASE and Cochrane databases for combination of terms "melatonin" and "delirium", restricted to clinical trials and up to October 25, 2017 found one relevant systematic review: this systematic review looked at the use of melatonin for delirium prevention and found four randomized control trials (RCT), out of which three showed positive results and one showed a negative result. Presently, despite its potential to reduce POD and improve sleep, the role of melatonin in the elderly surgical population is uncertain. There is a clear need for a large, well-designed study to establish definitive evidence.

ELIGIBILITY:
Inclusion Criteria:

* Age >65 years
* having a major non-cardiac surgery (which involve major vascular, thoracic, orthopedic, gynecological, otolaryngeal, general and gastrointestinal surgeries) with an expected hospital stay of 2 days or more, and
* ability to provide informed consent

Exclusion Criteria:

* active delirium or dementia
* ongoing melatonin treatment
* unable to take oral medications
* planned postoperative ventilation
* previous study participation
* allergy to melatonin
* hepatic impairment defined as alanine aminotransferase greater than 500 IU/L
* previous liver transplant or liver cirrhosis of Child-Pugh classes B and C
* not willing to participate
* language barrier

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2025-07-05 (Actual); Study Completion 2025-07-05 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 6 months
  Recruitment rate: assessed as at least 4-5 patients/week, and completion of recruitment (60 patients/site) in each site over 3-4 months.
Medication compliance | 8 days
  Proportion of patients who are able to take at least two doses of study medications, assessed as >85% of study patients.
Follow up to 3 months | 3 months
  Proportion of patients who complete 3 months follow up. For feasibility we expect >90% patients to complete study follow up.
Proportion of patients recruited from screening | 6 months
  To identify the proportion of screened patients meeting the study inclusion criteria

SECONDARY OUTCOMES:
Incidence of Delirium | 8 days
  This will be captured from observing the patient from the time of their discharge from pre-anesthetic care unit (PACU), until the time of discharge. Presence or absence will be captured using the Confusion Assessment Method (CAM)-short form. If patient is mechanically ventilated, the assessment will be performed using Confusion Assessment Method-Intensive Care Unit (CAM-ICU) tool.
Severity of Delirium | 8 days
  When an episode of post-operative delirium is observed, the severity will be assessed using Confusion Assessment Method (CAM) severity form. We will only record the severity for the first episode of post operative delirium observed.
Sleep quality | 8 days
  Quality of sleep will be assessed daily using Richards-Campbell Sleep Questionnaire (RCSQ). It is a visual analogue scale 0-100mm; zero indicating the worst possible sleep to 100 indicating the best sleep.
Incidence of ICU care | 8 days
  Need for ICU or critical care during hospitalization: This will be captured along with the reason and duration of such a stay from hospital records/patient charts
Prolonged hospital stay | 8 days
  Prolonged hospital stay (beyond anticipated for each patient) will be captured from hospital records/patient charts along with the reason and duration of such a stay
Institutional discharge | 3 months
  This will be recorded from hospital records.
Cognitive Status | 3 months
  This will be captured using Mini Mental Status Examination (MMSE)
Mortality | 3 months
  This outcome will be captured as in-hospital mortality and up to 3 months after discharge.
Adverse effects | 7 days
  Observe significant sedation using Pasero Opioid-induced Sedation Scale (validated, commonly used) S=Sleep, easy to arouse
  1. Awake and alert
  2. Slightly drowsy, easily aroused
     (S, 1, 2 all acceptable; no action necessary; may increase opioid dose if needed)
  3. Frequently drowsy, arousable, drifts off to sleep during conversation Unacceptable; monitor respiratory status and sedation level closely until sedation level is stable at <3 and respiratory status is satisfactory; decrease opioid dose 25% to 50%, or notifiy prescriber or anesthesiologist for orders; consider a non-sedation, opioid-sparing nonopioid if not contraindicated
  4. Somnolent, minimal or no response to verbal and physical stimulation Unacceptable; stop opioid; consider administering naloxone; notifiy prescriber or anesthesiologist; monitor respiratory status and sedation level closely until sedation level is stable at <3 and respiratory status is acceptable

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Hamilton Health Sciences-Juravinski Hospital Location, Hamilton, Ontario